CLINICAL TRIAL: NCT02736656
Title: Open-Label Extension Study to Evaluate the Long Term Safety and Efficacy of SPN-812 for the Treatment of Pediatric Patients With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Open-label Study to Evaluate Long-term Safety and Efficacy of SPN-812 (Viloxazine Extended-release Capsule)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812P310
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

ARMS (1):
- Open-Label Treatment (Experimental): Cohort 'A': Pediatric subjects 6-17 years of age who completed a Phase 2 (Study 812P202) or one of four Phase 3 trials (Study 812P301-P304).
  Cohort 'B': Pediatric subjects 4-5 years of age who completed a Phase 4 trial.
  Interventions: Drug: SPN-812

INTERVENTIONS:
Drug: SPN-812 — Cohort 'A': Children 6-11 yrs of age take 100-400mg SPN-812 once daily by mouth and adolescents 12-17 yrs of age take 100-600mg SPN-812 once daily by mouth. Pediatric subjects in Cohort 'A' are given a choice to extend their participation in the study every 6 months for up to 72 months.
  Cohort 'B': Pre-school-age children 4-5 yrs of age take 100mg SPN-812 once daily by mouth. Pediatric subjects in Cohort 'B' will be treated with 100 mg SPN-812 (100 mg capsule) for up to 6 months.
  Other Names: viloxazine extended-release capsules

SUMMARY:
Open label extension, long-term multicenter study of safety and efficacy of SPN-812 in pediatric ADHD patients

DETAILED DESCRIPTION:
This is a multicenter open-label extension study assessing long term safety and efficacy of SPN-812 (viloxazine extended-release capsules) in pediatric subjects with ADHD (A) who completed a Phase 2 (812P202: children 6 to 12 years of age) or one of four Phase 3 trials (812P301/812P303: children 6 to 11 years of age; 812P302/812P304: adolescents 12 to 17 years of age) or (B) who completed a Phase 4 trial (812P401: preschool-age children, 4-5 years of age). The study is divided into two phases, Optimization and Maintenance phases. Subjects in Cohort 'A' who completed a Phase 2 or Phase 3 trial followed protocol Schedule 'A' (exposure up to 72 months). Subjects in Cohort 'B' who complete the Phase 4 trial will follow Schedule 'B' (exposure up to 6 months).

ELIGIBILITY:
Cohort 'A' Inclusion/Exclusion Criteria:

Inclusion Criteria 'A':

1. Completion of a previous blinded study of SPN-812 for the treatment of ADHD.
2. Continues to be medically healthy and with clinically normal laboratory profiles, vital signs, and electrocardiograms (ECGs).
3. Weight of at least 20 kg if 6-11 years old and at least 35 kg if 12 years or older.
4. Written Informed Consent obtained from the subject's parent or legally authorized representative (LAR); and written Informed Assent obtained from the subject if appropriate; written Informed Consent obtained from the subject if he/she is 18 years old.
5. Females of Childbearing Potential (FOCP) must be either sexually inactive (abstinent) or, if sexually active, must agree to use one of the following acceptable birth control methods beginning 30 days prior to the first dose, throughout the study:

   1. simultaneous use of male condom and intra-uterine contraceptive device placed at least four weeks prior to the first study drug administration
   2. surgically sterile male partner
   3. simultaneous use of male condom and diaphragm with spermicide
   4. established hormonal contraceptive

Exclusion Criteria 'A':

1. Current diagnosis of significant systemic disease or of a major psychiatric or neurological disorder, including history or family history of seizures or seizure-like disorders. History of Major Depressive Disorder is allowed if the subject is free of episodes currently and for the last six months.
2. Current evidence of suicidal ideation and/or behaviors (assessed with Columbia Suicide Severity Rating Scale or C-SSRS).
3. Body Mass Index (BMI) greater than 95th percentile for the appropriate age and gender (according to the CDC BMI-for-Age Growth Charts for boys and girls).
4. Pregnancy, breastfeeding, or refusal to practice contraception during the study for female subjects of childbearing potential (FOCP).
5. Current substance or alcohol use.
6. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Cohort 'B' Inclusion/Exclusion Criteria:

Inclusion Criteria 'B':

1. Has completed a previous Study 812P401 and is less than 6 years of age at Visit 1 in this study (812P310).
2. Continues to be medically healthy with clinically normal laboratory profiles, vital signs, and electrocardiograms.
3. Weighs at least ≥5th percentile for age and sex.
4. Parent or LAR is willing and able to provide Written Informed Consent.

Exclusion Criteria 'B':

1. Has a current diagnosis of significant systemic disease and/or of a major psychiatric or neurological disorder.
2. Current evidence of suicidal ideation and/or behaviors (assessed with Columbia Suicide Severity Rating Scale or C-SSRS), is at significant risk of suicide, either in the opinion of the Investigator or defined as a "yes" to suicidal ideation C-SSRS questions 4 or 5 or answering "yes" to suicidal behavior on the C-SSRS at Visit 1 or has attempted suicide from day of end of study in previous blinded study to day of Visit 1 in this study (812P310).
3. Has a BMI >95th percentile for the appropriate age and sex (according to the CDC BMI-for-Age Growth Charts for boys and girls).
4. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1400 (Estimated)
Dates: Start 2016-02-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 72 months
  The incidence (percentage of subjects dosed) of adverse events by System Organ Class and Preferred term by cohort

SECONDARY OUTCOMES:
Trends in Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS-IV-Preschool, ADHD-RS-IV or ADHD-RS-5) Score | up to 72 months
  Change from Baseline in ADHD-RS Total score by visit by cohort
Trends in Clinical Global Impression-Improvement (CGI-I) scale score | up to 72 months
  CGI-I score by visit by cohort

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, MBA, Study Director — Supernus Pharmaceuticals, Inc.
Locations (16):
- United States (16):
  - Woodland International Research Group, Little Rock, Arkansas
  - Alliance for Wellness dba Alliance for Research, Long Beach, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Meridien Research at Florida Clinical Research Center, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Florida Clinical Research Center, LLC., Maitland, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - IPS Research, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - CNS Healthcare, Memphis, Tennessee
  - Bayou City Research Corporation, Houston, Texas
  - Road Runner Research, San Antonio, Texas
  - Ericksen Research & Development, Clinton, Utah
  - Northwest Clinical Trials, Bellevue, Washington

REFERENCES:
- [Derived] Findling RL, Katic A, Liebowitz M, Waxmonsky J, Fry N, Qin P, Yarullina I, Maldonado-Cruz Z, Lieberman VR, Rubin J. Viloxazine Extended-Release Capsules in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder: Results of a Long-Term, Phase 3, Open-Label Extension Trial. CNS Drugs. 2025 Nov;39(11):1157-1172. doi: 10.1007/s40263-025-01209-0. Epub 2025 Aug 13. PMID 40802027